CLINICAL TRIAL: NCT03779009
Title: Minimally INvasive Colon Cancer Surgery Through IMmunomics and Optical Mapping of the Sentinel Lymph Node.
Acronym: MINIMAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC/2017/1356
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colon Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tracer injection (Experimental)
  Interventions: Other: ICG-nanocoll (indocyanine green coupled to the human albumin colloidal particle nanocoll)

INTERVENTIONS:
Other: ICG-nanocoll (indocyanine green coupled to the human albumin colloidal particle nanocoll) — Under laparoscopic control, 2.0 ml of ICG-nanocoll will be injected into the subserosa at four quadrants around the tumor. Directly after injection, near infrared (NIR) fluorescence images (Olympus, Tokyo, Japan) will be acquired. SLNs will be identified and marked.

SUMMARY:
The project investigates the feasibility of laparoscopic fluorescent imaging for the intraoperative detection of the sentinel lymph node (SLN) in colon cancer patients. In addition, the topology of immunological and microenvironmental changes in normal and invaded lymph nodes (LN's) will be correlated to the LN location (anatomical mapping).

ELIGIBILITY:
Inclusion Criteria:

* Tumor type: proven adenocarcinoma of the colon
* Extent of disease (AJCC 7th edition): clinically node negative (stage II) non-metastatic colon cancer
* Locally resectable disease
* Adequate mental faculty, allowing to understand the proposed treatment protocol and provide informed consent
* Laboratory data

  * Serum creatinine ≤ 1.5 mg/dl or a calculated GFR ≥ 60 mL/min/1.73 m2
  * Serum total bilirubin ≤ 1.5 mg/dl, except for known Gilbert's disease
  * Platelet count > 100,000/µl
  * Hemoglobin > 9g/dl
  * Neutrophil granulocytes > 1,500/ml
  * International Normalized Ratio (INR) ≤ 2
* Absence of alcohol and/or drug abuse
* No inclusion in other clinical trials interfering with the study protocol
* No concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy
* Absence of any severe organ insufficiency
* No pregnancy or breast feeding
* Adequate contraception in fertile patients
* Written informed consent

Exclusion Criteria:

* Node positive and/or metastatic disease
* Locally unresectable disease
* Medically unfit patients (Karnofsky index < 70%)
* Allergies to any of the procedural substances (allergy to iodides, hypersensitivity to products containing human albumin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor status of the sentinel lymph node (SLN) and other lymph nodes (LN's) | up to 1 month after surgery
  All LN in the resection specimen will be collected, mapped, and labeled. The SLN is defined as fluorescent hotspot that appears after injection of the tracer. Standard H&E staining will be performed on LN sections and all mapped LN (including the SLN) will be analyzed for their tumor status.

SECONDARY OUTCOMES:
Immunological markers | up to 12 months after surgery
  Single cell suspensions will be prepared from all LN (including the SLNs) and the primary tumor. Cell suspensions will be analyzed for cytotoxic CD8+ CD45RO+T cells, CD4+ T helper cells, dendritic cell subsets (DC), natural killer (NK) cells, tumor-associated macrophages (TAM), and myeloid-derived suppressor cells (MDSCs) by multicolor fluorescence-activated cell sorting (FACS)-based immuno-panels. FACS is technique to detect and measure physical and chemical characteristics of a population of cells and provides quantifiable data.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No